CLINICAL TRIAL: NCT02776748
Title: An Open-label, Short-duration, Repeat-dose Study of Breastmilk Excretion and Infant Absorption of Daily Oral Tenofovir Disoproxil Fumarate/Emtricitabine When Used by HIV-uninfected Lactating Women
Brief Title: PrEP in Breastfeeding Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Jared Baeten, Professor, Global Health, Medicine, & Epidemiology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 46363
Record Dates: First submitted 2016-05-15; First posted 2016-05-18 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: HIV Pre-exposure Prophylaxis During Breastfeeding
Keywords: Tenofovir disoproxil; Pre-exposure prophylaxis; Breastfeeding; Emtricitabine; Tenofovir; Post-partum; HIV prevention; Women; Pharmacokinetics
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FTC-TDF (Other): Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) PrEP: 200mg FTC /300 mg TDF
  Interventions: Drug: FTC/TDF PrEP

INTERVENTIONS:
Drug: FTC/TDF PrEP — Daily oral directly observed FTC/TDF PrEP administered to breastfeeding HIV-uninfected women
  Other Names: Truvada PrEP

SUMMARY:
The purpose of this study is to quantify the magnitude and extent of infant exposure to daily emtricitabine (FTC) /tenofovir disoproxil fumarate (TDF) via maternal breastmilk when taken pre-exposure prophylaxis (PrEP) by lactating HIV-uninfected women. The primary outcome is the steady state concentrations of emtricitabine and tenofovir in the infant plasma.

DETAILED DESCRIPTION:
This is prospective, short-duration, open-label, single-arm, repeat-dose, pharmacokinetic study of daily FTC/TDF PrEP among HIV-uninfected lactating mother-infant pairs. PrEP will be administered to women through daily directly observed therapy for 10 consecutive days - sufficient to reach steady-state but discontinuing thereafter. No drug will be administered to the infant directly. Co-formulated FTC and TDF were dosed at 200 mg daily and 300 mg daily, respectively. The overall goal is to quantify the magnitude and degree to which breastfeeding infants are exposed to FTC/TDF when used as PrEP by HIV-uninfected lactating women. Maternal blood and breastmilk samples will be obtained concurrently (i.e., within 30 minutes of each other) regardless of the timing of food intake (i.e., non-fasting) on the 7th and 10th day. Peak samples will be obtained 1-2 hours after the maternal directly observed PrEP and trough samples were obtained at the end of the dosing interval (i.e., 23 to 24 hours after directly observed PrEP dose). A single infant blood sample will be obtained after the maternal 7th directly observed PrEP dose.

We will conduct quantitative measurements and analyses of infant plasma drug concentrations, infant-plasma to breastmilk and breastmilk to maternal plasma drug concentration ratios to characterize FTC and TDF transmission to breast feeding infants. Tenofovir and emtricitabine concentrations in plasma and breastmilk will be quantified via previously validated liquid chromatographic-tandem mass spectrometric (LC-MS/MS) methods in accordance with the recommendations included in the US Food and Drug Administration, Guidance for Industry, Bioanalytical Method Validation guidelines.

ELIGIBILITY:
Inclusion Criteria:

For infant's mother and father

* Able and willing to provide informed consent for the infant to participate in the study
* Of legal age ≥18 years to consent

For HIV-uninfected mother, in addition to the criteria noted immediately above:

* Willing to provide breast milk samples and breastfeed during the duration of the study 0-24 weeks postpartum
* Breastfeeding an infant
* HIV-uninfected based on negative HIV rapid tests, both at study screening and at the enrollment visit
* Adequate renal function, defined by normal creatinine levels and estimated creatinine clearance ≥60 mL/min
* Not infected with hepatitis B virus, as determined by a negative hepatitis B surface antigen test
* Not currently using PrEP
* Note: single mothers will be eligible to participate in this study. Where possible the father's permission was be obtained. When the father is unknown, incompetent, deceased, or not reasonably available, or when only the mother has the legal responsibility for the care and custody of the child, infant participation will be based on the mother's consent and documentation will be added to file.

For infant

* Infant born to eligible women (both male and female infants will be included)
* Age 0-24 weeks
* Otherwise infant has no serious infections or active clinically significant medical problems

Exclusion Criteria:

* Women breastfeeding more than one child
* Preterm babies or infants with low birth weight (i.e. ≤2000mg)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Steady state plasma concentrations of emtricitabine and tenofovir in the infants of breastfeeding women using PrEP: Quantity of PrEP medications in the infant plasma. | Time averaged: 10 days
  Infant exposure measured as median (interquartile range) concentrations of emtricitabine and tenofovir infant plasma.
Steady state plasma concentrations of emtricitabine and tenofovir in the infants of breastfeeding women using PrEP: Detectable and quantifiable concentrations of PrEP medications in the infant plasma. | Time averaged: 10 days
  Measure the proportion of infant plasma samples with concentrations of emtricitabine and tenofovir below the assay lower limit of quantification.
Steady state concentrations of emtricitabine and tenofovir in plasma of HIV-uninfected women using PrEP. | Time averaged: 10 days
  Measure median (interquartile range) concentrations of emtricitabine and tenofovir in maternal plasma.
Steady state concentrations of emtricitabine and tenofovir in breastmilk of HIV-uninfected women using PrEP. | Time averaged: 10 days
  Measure median (interquartile range) concentrations of emtricitabine and tenofovir in breast milk.
Infant plasma-to-maternal breast milk emtricitabine and tenofovir concentration ratios. | Time averaged: 10 days
  Measure median (interquartile range) infant plasma-to-maternal breast milk emtricitabine and tenofovir concentration ratios.
Infant daily dose of tenofovir and emtricitabine received from breastmilk | Time averaged: 10 days
  We will compute the infant drug dose received from breastmilk per day (infant Computed as the product of breast milk tenofovir and emtricitabine concentrations and the estimated volume of breast milk consumed by infant daily. We will assume the daily amount of breast milk consumed by the infant to be 150 mL/kg/day, the standardized milk consumption of the average milk intake of a fully breast-fed infant. Measure median (interquartile range) infant daily dose for tenofovir and emtricitabine from breastmilk.
Infant dose fraction for tenofovir and emtricitabine. | Time averaged: 10 days
  Infant dose fraction (i.e., exposure index) represents the daily amount of drug dose an infant would ingest from breast milk as a percentage of the recommended pediatric therapeutic daily dose. Infant dose fraction will be computed as as: infant dose fraction (%) = infant dose from breast milk *100/infant therapeutic dose. Measure median (interquartile range) infant dose fraction.
Maternal breastmilk emtricitabine and tenofovir to plasma concentration ratios. | Time averaged: 10 days
  Measure median (interquartile range) of maternal breastmilk emtricitabine and tenofovir to plasma concentration ratios.
Serious adverse events in infants of breastfeeding HIV-uninfected women using PrEP. | Time averaged: 10 days
  Number of infants with serious adverse effects.
Serious adverse events in breastfeeding HIV-uninfected women using PrEP. | Time averaged: 10 days
  Number of women with serious adverse effects.

CONTACTS AND LOCATIONS:
Overall Officials: Jared M Baeten, MD, PhD, Principal Investigator — University of Washington; Kenneth K Mugwanya, MBChB, MS, Study Director — University of Washington
Locations (2):
- Partners in Prevention-Thika, Thika, Kenya
- Partners in Prevention-Infectious Diseases Institute LTD, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Data from the PrEP in Breastfeeding Study are available by contacting the International Clinical Research Center at the University of Washington (icrc@uw.edu).

REFERENCES:
- [Derived] Mugwanya KK, Hendrix CW, Mugo NR, Marzinke M, Katabira ET, Ngure K, Semiyaga NB, John-Stewart G, Muwonge TR, Muthuri G, Stergachis A, Celum CL, Baeten JM. Pre-exposure Prophylaxis Use by Breastfeeding HIV-Uninfected Women: A Prospective Short-Term Study of Antiretroviral Excretion in Breast Milk and Infant Absorption. PLoS Med. 2016 Sep 27;13(9):e1002132. doi: 10.1371/journal.pmed.1002132. eCollection 2016 Sep. PMID 27676257